CLINICAL TRIAL: NCT03627871
Title: Enduring Exercise Habits: Trending Norms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 827107-1237
Record Dates: First submitted 2018-08-02; First posted 2018-08-14 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: exercise; social norms; interest in exercising more
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Trending majority norm (Experimental): Participants receive information about exercise-related norms that apply to the majority of the population and are told this norm has been increasing recently.
  Interventions: Behavioral: Trending Majority Norm
- Non-trending majority norm (Experimental): Participants receive information about exercise-related norms that apply to the majority of the population but are not told about recent trends.
  Interventions: Behavioral: Majority Norm
- Trending minority norm (Experimental): Participants receive information about exercise-related norms that apply to a minority of the population and are told this norm has been increasing recently
  Interventions: Behavioral: Trending Minority Norm
- Non-trending minority norm (Experimental): Participants receive information about exercise-related norms that apply to a minority of the population but are not told about recent trends.
  Interventions: Behavioral: Minority Norm
- Control (Experimental): Participants receive information about exercise unrelated to social norms or recent trends.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Majority Norm — Participants receive information about exercise norms that apply to the majority of the population but are given no information about trends in this norm.
  Arms: Non-trending majority norm
Behavioral: Trending Minority Norm — Participants receive information about exercise norms that apply to the minority of the population and have recently been trending up.
  Arms: Trending minority norm
Behavioral: Minority Norm — Participants receive information about exercise norms that apply to the minority of the population but are given no information about trends in this norm.
  Arms: Non-trending minority norm
Behavioral: Control — Participants receive information about exercise that is unrelated to social norms or trends in social norms.
  Arms: Control
Behavioral: Trending Majority Norm — Participants receive information about exercise norms that apply to the majority of the population and have recently been trending up.
  Arms: Trending majority norm

SUMMARY:
Learning that most people engage in an activity can be a powerful motivator to adoption. But are there instances in which people can similarly find motivation from learning that only a minority of others engage in a behavior? Evidence suggests this may be possible when the message is that the size of the minority has been growing in recent years. In this study, we first examine how gym members' exercise patterns shift when they are informed that the minority versus the majority of (a subpopulation of) other Americans exercise frequently. We also test how gym members are affected by learning that the number of frequent exercisers has increased in recent years.

DETAILED DESCRIPTION:
Gym members register online to participate in a 28-day workout program. Upon registration, participants are assigned to one of five conditions (a 2 x 2 study design plus a control group). Participants are assigned to receive information about majority exercise norms or minority exercise norms, and are informed that these norms are trending up or receive no information about trends in these norms. Participants are then prompted to create a workout schedule. Over the 28-day intervention period, participants are sent text messages with information about exercise depending on their condition (i.e., majority trending exercise norms, majority exercise norms with no information about trends, minority trending exercise norms or minority norms with no information about trends), workout reminders before their scheduled workouts, and weekly emails with additional exercise information related to their assigned condition and their schedule. Participants assigned to the control condition are prompted to create a workout schedule and receive text message reminders, information about exercise that is unrelated to social norms, and weekly emails with exercise information unrelated to social norms or trends and their workout schedule. All participants earn points for participating and for each day that they go to the gym which can be redeemed for an Amazon cash gift card after the end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Has 24 Hour Fitness gym membership

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Gym visits per week | During the 28-day intervention period
  Number of times the participant goes to the gym
Gym visits per week | During the 4-weeks post-intervention
  Number of times the participant goes to the gym
Gym visits per week | During the 10-weeks post-intervention
  Number of times the participant goes to the gym
Whether or not a participant visits the gym in a given week | During the 28-day intervention period
  Binary variable capturing whether or not a participant had any gym visits in a given week
Whether or not a participant visits the gym in a given week | During the 4-weeks post-intervention
  Binary variable capturing whether or not a participant had any gym visits in a given week
Whether or not a participant visits the gym in a given week | During the 10-weeks post-intervention
  Binary variable capturing whether or not a participant had any gym visits in a given week

SECONDARY OUTCOMES:
Gym visits per week | During the 52-weeks post-intervention
  Number of times the participant goes to the gym
Whether or not a participant visits the gym in a given week | During the 52-weeks post-intervention
  Binary variable capturing whether or not a participant had any gym visits in a given week

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No